CLINICAL TRIAL: NCT02809768
Title: A 3-Part, Open-Label Study to Assess Pharmacokinetic Drug-Drug Interaction Between Avatrombopag When Co-Administered With Fluconazole (Moderate Inhibitor of CYP2C9 and CYP3A), Itraconazole (Strong CYP3A Inhibitor), or Rifampin (Strong CYP3A and Moderate CYP2C9 Inducer) in Healthy Subjects
Brief Title: Study to Assess Pharmacokinetic Drug-Drug Interaction Between Avatrombopag When Co-Administered With Fluconazole, Itraconazole, or Rifampin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E5501-A001-019
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Healthy Participants
Keywords: Healthy participants; Pharmacokinetic Drug-Drug Interaction; Avatrombopag
MeSH Terms: interventions — avatrombopag; Fluconazole; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Avatrombopag plus fluconazole (Experimental): Part A: Participants will be administered a single oral dose of avatrombopag (20-mg) on Day 1 of Treatment Period 1. In Treatment Period 2, fluconazole (400-mg) will be administered once daily on Days 1 to 16, and a single dose of avatrombopag (20-mg) on Day 7 in Treatment Period 2. Each dose of avatrombopag will be administered under fed conditions 30 minutes after the start of a meal.
  Interventions: Drug: Avatrombopag; Drug: Fluconazole
- Avatrombopag plus itraconazole (Experimental): Part B: Participants will be administered a single oral dose of avatrombopag (20-mg) on Day 1 of Treatment Period 1. In Treatment Period 2, itraconazole (200-mg) will be administered twice daily on Day 1 and 200-mg once daily on Days 2 to 16. A single dose of avatrombopag (20-mg) will be administered on Day 7 of Treatment Period 2. Each dose of avatrombopag will be administered under fed conditions 30 minutes after the start of a meal.
  Interventions: Drug: Avatrombopag; Drug: Itraconazole
- Avatrombopag plus rifampin (Experimental): Part C: Participants will be administered a single oral dose of avatrombopag (20-mg) on Day 1 of Treatment Period 1. In Treatment Period 2, rifampin (600-mg) will be administered once daily on Days 1 to 16. In order to avoid a food-effect on rifampin absorption, each dose will be administered 1 hour before participants consume a meal. On Day 7 of Treatment Period 2, rifampin (600-mg) and avatrombopag (20-mg) will be administered 1 hour before meal and 30 minutes after starting meal consumption.
  Interventions: Drug: Avatrombopag; Drug: Rifampin

INTERVENTIONS:
Drug: Avatrombopag
  Other Names: E5501
Drug: Fluconazole
  Arms: Avatrombopag plus fluconazole
Drug: Itraconazole
  Arms: Avatrombopag plus itraconazole
Drug: Rifampin
  Arms: Avatrombopag plus rifampin

SUMMARY:
The purpose of this study is to determine the effects of concomitant administration with fluconazole, itraconazole, and rifampin on the pharmacokinetics (PK) of a single 20-mg dose of avatrombopag in healthy participants.

DETAILED DESCRIPTION:
This study will be a single center, open-label, drug-drug interaction study in healthy participants. The study will consist of 3 parts: In Part A, the effects of steady-state dosing of a moderate inhibitor of CYP2C9 and CYP3A (fluconazole) on the single-dose PK of avatrombopag will be assessed. In Part B, the effects of steady-state dosing of a strong CYP3A inhibitor (itraconazole) on the single-dose PK of avatrombopag will be assessed. In Part C, the effects of steady-state dosing of a strong CYP3A and moderate CYP2C9 inducer (rifampin) on the single-dose PK of avatrombopag will be assessed.

Each Part of the study will consist of 2 phases: Pretreatment and Treatment. The Pretreatment Phase will consist of 2 periods: Screening and Baseline Period 1.The Treatment Phase will consist of 2 treatment periods: Treatment Period 1 (administration of a single oral dose of avatrombopag 20 mg alone under fed conditions); and Treatment Period 2 (administration of oral doses of each inhibitor or inducer alone and concomitant administration of a single oral dose of avatrombopag 20 mg with each inhibitor or inducer [fluconazole in Part A, itraconazole in Part B, or rifampin in Part C] under fed conditions).

ELIGIBILITY:
Inclusion Criteria:

1. Platelet count between the lower limit of normal and 300 × 10^9/L, inclusive, at Screening and each Baseline.
2. Non-smoking, male or female, age ≥18 years and ≤55 years old.
3. Body mass index (BMI) >18 and ≤32 kg/m^2 at Screening.
4. Females must not be pregnant at Screening as documented by a negative serum beta human chorionic gonadotropin (β-hCG) test with a minimum sensitivity 25 IU/L or equivalent units of β-hCG or at Baseline as documented by a negative urine pregnancy test result.

Exclusion Criteria:

1. Failure to discontinue use of agents associated with higher risk of thrombosis (including estrogen containing oral contraceptives) within at least 30 days before dosing.
2. Evidence of organ dysfunction or any clinically significant deviation from normal in their medical history (e.g., history of splenectomy); history of arterial or venous thrombosis, including partial or complete thromboses (e.g., stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis, pulmonary embolism); known family history of hereditary thrombophilic disorders (e.g., Factor V Leiden, antithrombin III deficiency).
3. Hemoglobin less than lower limit of normal at Screening and Baseline Period 1.
4. Liver functions tests (alanine transaminase [ALT], aspartate transaminase [AST], or total bilirubin) greater than the upper limit of normal Screening and Baseline Period 1.
5. Any history of gastrointestinal surgery that may affect the pharmacokinetics (PK) profiles of avatrombopag (e.g., hepatectomy, nephrectomy, cholecystectomy or digestive organ resection) at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mean maximum observed concentration (Cmax) | Predose of Day 1 (Treatment Period 1), Predose of Day 7 (Treatment Period 2), and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 144, and 216 hours postdose of avatromobag for Treatment period 1 and 2
Median time at which the highest drug concentration occurs (tmax) | Predose of Day 1 (Treatment Period 1), Predose of Day 7 (Treatment Period 2), and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 144, and 216 hours postdose of avatromobag for Treatment period 1 and 2
Mean area under the concentration-time curve from zero time to time of last quantifiable concentration AUC(0-t) | Predose of Day 1 (Treatment Period 1), Predose of Day 7 (Treatment Period 2), and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 144, and 216 hours postdose of avatromobag for Treatment period 1 and 2
Mean area under the concentration-time curve from zero time to 72 hours postdose AUC(0-72h) | Predose of Day 1 (Treatment Period 1), Predose of Day 7 (Treatment Period 2), and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 144, and 216 hours postdose of avatromobag for Treatment period 1 and 2
Mean terminal elimination phase half-life (t1/2) | Predose of Day 1 (Treatment Period 1), Predose of Day 7 (Treatment Period 2), and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 144, and 216 hours postdose of avatromobag for Treatment period 1 and 2
Mean apparent total clearance following oral administration (CL/F) | Predose of Day 1 (Treatment Period 1), Predose of Day 7 (Treatment Period 2), and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 144, and 216 hours postdose of avatromobag for Treatment period 1 and 2
Mean apparent volume of distribution at terminal phase (Vz/F) | Predose of Day 1 (Treatment Period 1), Predose of Day 7 (Treatment Period 2), and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 144, and 216 hours postdose of avatromobag for Treatment period 1 and 2
Mean area under the concentration-time curve from zero time extrapolated to infinite time AUC(0-inf) | Predose of Day 1 (Treatment Period 1), Predose of Day 7 (Treatment Period 2), and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72, 96, 144, and 216 hours postdose of avatromobag for Treatment period 1 and 2

SECONDARY OUTCOMES:
Mean maximum platelet counts following avatrombopag dosing observed in each treatment period (Emax) | Predose of Day 1, Days 3, 4, 5, 7, 10, 12, 14, 21, and 28 of Treatment Period 1. Predose of Day 7, Days 9, 10, 11, 13, 16, 18, 20, 27, and 34 of Treatment Period 2
Median observed time of maximum increase in platelet counts following avatrombopag dosing in each treatment period (TEmax) | Predose of Day 1, Days 3, 4, 5, 7, 10, 12, 14, 21, and 28 of Treatment Period 1. Predose of Day 7, Days 9, 10, 11, 13, 16, 18, 20, 27, and 34 of Treatment Period 2
Mean area under the effect curve for platelet count following avatrombopag dosing through 28 days after dosing (AUEC(0-28d)) | Predose of Day 1, Days 3, 4, 5, 7, 10, 12, 14, 21, and 28 of Treatment Period 1. Predose of Day 7, Days 9, 10, 11, 13, 16, 18, 20, 27, and 34 of Treatment Period 2
Maximum change from baseline in platelet count (ΔEmax = Emax - baseline platelet count at predose on Treatment Period 1 Day 1) (ΔEmax) | Predose of Day 1, Days 3, 4, 5, 7, 10, 12, 14, 21, and 28 of Treatment Period 1. Predose of Day 7, Days 9, 10, 11, 13, 16, 18, 20, 27, and 34 of Treatment Period 2
Maximum percent change from baseline in platelet count (%ΔEmax = ΔEmax / baseline platelet count at predose on Period 1 Day 1 x 100) (%ΔEmax) | Predose of Day 1, Days 3, 4, 5, 7, 10, 12, 14, 21, and 28 of Treatment Period 1. Predose of Day 7, Days 9, 10, 11, 13, 16, 18, 20, 27, and 34 of Treatment Period 2
Percentage of participants with treatment emergent adverse events and serious adverse events | Up to approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Information, Study Director — Eisai Inc.
Locations (1):
- San Antonio, Texas, United States